CLINICAL TRIAL: NCT01425008
Title: An Open-Label, Phase 1, Dose Escalation Study of MLN2480 in Patients With Relapsed or Refractory Solid Tumors Followed by a Dose Expansion Phase in Patients With Metastatic Melanoma
Brief Title: Study of MLN2480 in Participants With Relapsed or Refractory Solid Tumors Followed by a Dose Expansion in Participants With Metastatic Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C28001; 2012-003397-16 (EudraCT Number); U1111-1164-7508 (Registry Identifier: WHO); 13/SC/0007 (Registry Identifier: NRES)
Record Dates: First submitted 2011-08-26; First posted 2011-08-29 (Estimated); Results first posted 2020-08-10 (Actual); Last update posted 2020-08-10 (Actual); Status verified 2020-07

CONDITIONS: Melanoma; Metastatic Melanoma; Solid Tumor; Neoplasm
Keywords: Drug Therapy
MeSH Terms: conditions — Melanoma; Neoplasms | interventions — tovorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MLN2480 (Experimental)
  Interventions: Drug: MLN2480

INTERVENTIONS:
Drug: MLN2480 — Dose Escalation Phase: participants will receive MLN2480 orally in escalating doses every other day or once weekly for three weeks of a 28-day cycle. Participants may continue treatment for additional cycles (up to 12 months) until disease progression, unacceptable toxicity, or the participant discontinues for any other reason. If it is determined that a participant would derive benefit from continued therapy beyond 12 months treatment may continue. Dose Expansion Phase: Participants will take MLN2480 at the maximum tolerated dose orally every other day or once weekly for three weeks of a 28-day cycle until disease progression, unacceptable toxicity, or the participant discontinues for any other reason. The maximum duration of treatment is 1 year unless determined that a participant would derive benefit from continued therapy beyond 12 months.
  Other Names: TAK-580

SUMMARY:
This is a phase 1, multicenter, nonrandomized, open-label, dose escalation study. The study will be conducted in 2 stages, Dose Escalation and Dose Expansion. The Dose Escalation phase will include participants with solid tumors (including melanoma) who have failed or are not candidates for standard therapies or for whom no approved therapy is available. The Dose Expansion phase will include participants with metastatic melanoma.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent.
2. Male or female participants 18 years or older.
3. Dose Escalation phase: Participants with solid tumors (including melanoma) who have failed or are not candidates for standard therapies of for whom no approved therapy is available.
4. Dose Expansion phase: Metastatic melanoma (locally advanced or metastatic melanoma).
5. Dose Expansion phase: At least 1 measurable lesion which has not been treated previously with radiotherapy. A newly arising lesion in a previously irradiated field is acceptable.
6. For participants undergoing biopsy procedures: Prothrombin time (PT) and activated partial thromboplastin time (aPTT) must be within the normal range.
7. Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to (<=) 1.
8. Adequate tissue sample from either archival formalin-fixed paraffin-embedded (FFPE) tumor tissue or new biopsy of tumor.
9. Previous chemotherapy, immunotherapy, and hormone therapy must be completed at least 4 weeks prior to the administration of MLN2480 and radiation must be completed at least 3 weeks prior to the administration of MLN2480; all associated toxicity must be resolved to <=Grade 1.
10. Expected survival time of at least 3 months in the opinion of the investigator.
11. Participants who do not have hypo- or hyperthyroidism.
12. Ability to swallow and retain oral medication.
13. Female participants who are postmenopausal for at least 1 year, surgically sterile, or agree to practice 2 effective methods of contraception through 3 months after the last dose of study drug or agree to practice true abstinence.
14. Male participants who, even if surgically sterilized, agree to practice effective barrier contraception through 3 months after the last dose of alisertib or agree to practice true abstinence.

Exclusion Criteria

1. History of any major disease that might interfere with safe protocol participation.
2. Dose Expansion phase: Previous treatment with RAF or MEK inhibitors.
3. Laboratory values as specified in study protocol.
4. Current enrollment in any other investigational treatment study.
5. Evidence of current uncontrolled cardiovascular conditions within the past 6 months.
6. Prior investigational agents for malignant or non-malignant disease within 4 weeks prior to Day 1.
7. Active hepatitis or human immunodeficiency virus (HIV) infection.
8. Active bacterial or viral infection.
9. Female participants who are pregnant or currently breastfeeding.
10. Major surgery within 28 days of Day 1.
11. Refractory nausea and vomiting, malabsorption, or significant bowel or stomach resection.
12. Inability to comply with study requirements.
13. Other unspecified reasons that, in the opinion of the investigator or Millennium, make the participant unsuitable for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2011-09-15 (Actual); Primary Completion 2017-04-11 (Actual); Study Completion 2018-10-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.
Locations (16):
- United States (9):
  - San Francisco, California
  - Denver, Colorado
  - Augusta, Georgia
  - Indianapolis, Indiana
  - New York, New York
  - Easton, Pennsylvania
  - Philadelphia, Pennsylvania
  - San Antonio, Texas
  - Lakewood, Washington
- United Kingdom (7):
  - Bristol, Avon
  - Cambridge, Cambridgeshire
  - Chelmsford, Essex
  - London, Greater London
  - Manchester, Greater Manchester
  - Oxford, Oxfordshire
  - Newcastle upon Tyne, Tyne & Wear

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment."

REFERENCES:
- [Derived] Rasco DW, Medina T, Corrie P, Pavlick AC, Middleton MR, Lorigan P, Hebert C, Plummer R, Larkin J, Agarwala SS, Daud AI, Qiu J, Bozon V, Kneissl M, Barry E, Olszanski AJ. Phase 1 study of the pan-RAF inhibitor tovorafenib in patients with advanced solid tumors followed by dose expansion in patients with metastatic melanoma. Cancer Chemother Pharmacol. 2023 Jul;92(1):15-28. doi: 10.1007/s00280-023-04544-5. Epub 2023 May 23. PMID 37219686

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 16 investigative sites in the United States and United Kingdom from 13 September 2011 to 16 October 2018.
Pre-assignment Details: Participants with relapsed and refractory solid tumors and metastatic melanoma were enrolled in Dose Escalation Phase and Dose Expansion Phase respectively to receive TAK-580 (MLN2480), once every other day (Q2D) or once weekly (QW). Q2D Dose Expansion Phase, TAK-580 (BRAF+) was discontinued due to sponsor's decision of strategic deprioritization.
Groups:
- Q2D Dose Escalation Phase: TAK-580 20 mg (22 Days Cycle): TAK-580 20 milligram (mg), tablets, orally, Q2D, in each 22-days treatment cycle until disease progression, unacceptable toxicity, or participant discontinuation for any other reason (up to Cycle 38).
- Q2D Dose Escalation Phase: TAK-580 40 mg (22 Days Cycle): TAK-580 40 mg, tablets, orally, Q2D, in each 22-days treatment cycle until disease progression, unacceptable toxicity, or participant discontinuation for any other reason (up to Cycle 38).
- Q2D Dose Escalation Phase: TAK-580 80 mg (22 Days Cycle): TAK-580 80 mg, tablets, orally, Q2D, in each 22-days treatment cycle until disease progression, unacceptable toxicity, or participant discontinuation for any other reason (up to Cycle 38).
- Q2D Dose Escalation Phase: TAK-580 135 mg (22 Days Cycle): TAK-580 135 mg, tablets, orally, Q2D, in each 22-days treatment cycle until disease progression, unacceptable toxicity, or participant discontinuation for any other reason (up to Cycle 38).
- Q2D Dose Escalation Phase: TAK-580 200 mg (22 Days Cycle): TAK-580 200 mg, tablets, orally, Q2D, in each 22-days treatment cycle until disease progression, unacceptable toxicity, or participant discontinuation for any other reason (up to Cycle 38).
- Q2D Dose Escalation Phase: TAK-580 280 mg (22 Days Cycle): TAK-580 280 mg, tablets, orally, Q2D, in each 22-days treatment cycle until disease progression, unacceptable toxicity, or participant discontinuation for any other reason (up to Cycle 38).
- Q2D Dose Escalation Phase: TAK-580 200 mg (28 Days Cycle): TAK-580 200 mg, tablets, orally, Q2D, in each 28-days treatment cycle until disease progression, unacceptable toxicity, or participant discontinuation for any other reason (up to Cycle 38).
- QW Dose Escalation Phase: TAK-580 400 mg (28 Days Cycle): TAK-580 400 mg, tablets, orally, QW, in each 28-days treatment cycle until disease progression, unacceptable toxicity, or participant discontinuation for any other reason (up to Cycle 38).
- QW Dose Escalation Phase: TAK-580 600 mg (28 Days Cycle): TAK-580 600 mg, tablets, orally, QW, in each 28-days treatment cycle until disease progression, unacceptable toxicity, or participant discontinuation for any other reason (up to Cycle 38).
- QW Dose Escalation Phase: TAK-580 800 mg (28 Days Cycle): TAK-580 800 mg, tablets, orally, QW, in each 28-days treatment cycle until disease progression, unacceptable toxicity, or participant discontinuation for any other reason (up to Cycle 38).
- Q2D Dose Expansion Phase: TAK-580 (BRAF+ Naive): TAK-580 200 mg, tablets, orally, Q2D, in each 28-days treatment cycle until disease progression, unacceptable toxicity, or participant discontinuation for any other reason (up to Cycle 49) in participants with BRAF mutation-positive cutaneous melanoma, naive to prior therapy with rapidly accelerated fibrosarcoma (RAF) and mitogen-activated protein kinase (MEPK kinase) or extracellular signal-regulated kinase (ERK kinase) (MEK) inhibitors.
- Q2D Dose Expansion Phase: TAK-580 (BRAF+ Previously Treated): TAK-580 200 mg, tablets, orally, Q2D, in each 28-days treatment cycle until disease progression, unacceptable toxicity, or participant discontinuation for any other reason (up to Cycle 49) in participants with BRAF mutation-positive cutaneous melanoma, which in response to previous treatment with RAF inhibitors and/or MEK inhibitors had relapsed following an objective response, failed to demonstrate an objective response and/or could not tolerate such a regimen due to unacceptable toxicity.
- Q2D Dose Expansion Phase: TAK-580 (NRAS+ Naive): TAK-580 200 mg, tablets, orally, Q2D, in each 28-days treatment cycle until disease progression, unacceptable toxicity, or participant discontinuation for any other reason (up to Cycle 49) in participants with NRAS mutation-positive cutaneous melanoma, naive to prior therapy with RAF and MEK inhibitors.
- Q2D Dose Expansion Phase: TAK-580 (NRAS+ Previously Treated): TAK-580 200 mg, tablets, orally, Q2D, in each 28-days treatment cycle until disease progression, unacceptable toxicity, or participant discontinuation for any other reason (up to Cycle 49) in participants with NRAS mutation-positive cutaneous melanoma, which in response to previous treatment with MEK inhibitors had relapsed following an objective response, failed to demonstrate an objective response and/or could not tolerate such a regimen due to unacceptable toxicity.
- Q2D Dose Expansion Phase: TAK-580 BRAF/NRAS WT+ Naive: TAK-580 200 mg, tablets, orally, Q2D, in each 28-days treatment cycle until disease progression, unacceptable toxicity, or participant discontinuation for any other reason (up to Cycle 49) in participants with BRAF/NRAS mutation-negative cutaneous melanoma (wild type [WT]), naive to any prior anticancer therapy except ipilimumab, anti-programmed cell death-1 (PD-1), and anti-PD ligand-1 (PDL-1) monoclonal antibodies.
- Q2D Dose Expansion Phase:TAK-580 BRAF/NRASWT+PreviouslyTreated: TAK-580 200 mg, tablets, orally, Q2D, in each 28-days treatment cycle until disease progression, unacceptable toxicity, or participant discontinuation for any other reason (up to Cycle 49) in participants with BRAF/NRAS mutation-negative melanoma (WT), who had received at least 1 line of prior anticancer therapy.
- Q2D Dose Expansion Phase: Pharmacokinetic Cohort: TAK-580 200 mg, tablets, orally, on Days 1 through 21 in a 28-days treatment Cycle 1, followed by TAK-580 200 mg, tablets, orally, Q2D in each 28-days treatment cycle from Cycle 2 until disease progression, unacceptable toxicity, or participant discontinuation for any other reason (up to Cycle 49) in participants with any advanced solid tumor (excluding lymphoma, but including melanoma) who had failed or were not candidates for standard therapies or for whom no approved therapy was available.
- Q2D Dose Expansion Phase: TAK-580 (BRAF+): TAK-580 200 mg, tablets, orally, Q2D, in each 28-days treatment cycle until disease progression, unacceptable toxicity, or participant discontinuation for any other reason (up to Cycle 49) in participants with BRAF-mutation positive cutaneous melanoma.
- QW Dose Expansion Phase: TAK-580 NRAS WT+ Naive: TAK-580 600 mg, tablets, orally, QW, in each 28-days treatment cycle until disease progression, unacceptable toxicity, or participant discontinuation for any other reason (up to Cycle 49), in participants with NRAS mutation-positive cutaneous melanoma, naive to prior therapy with RAF and MEK inhibitors.
Period: Dose Escalation Phase
Arm/Group | Q2D Dose Escalation Phase: TAK-580 20 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 40 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 80 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 135 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 200 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 280 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 200 mg (28 Days Cycle) | QW Dose Escalation Phase: TAK-580 400 mg (28 Days Cycle) | QW Dose Escalation Phase: TAK-580 600 mg (28 Days Cycle) | QW Dose Escalation Phase: TAK-580 800 mg (28 Days Cycle) | Q2D Dose Expansion Phase: TAK-580 (BRAF+ Naive) | Q2D Dose Expansion Phase: TAK-580 (BRAF+ Previously Treated) | Q2D Dose Expansion Phase: TAK-580 (NRAS+ Naive) | Q2D Dose Expansion Phase: TAK-580 (NRAS+ Previously Treated) | Q2D Dose Expansion Phase: TAK-580 BRAF/NRAS WT+ Naive | Q2D Dose Expansion Phase:TAK-580 BRAF/NRASWT+PreviouslyTreated | Q2D Dose Expansion Phase: Pharmacokinetic Cohort | Q2D Dose Expansion Phase: TAK-580 (BRAF+) | QW Dose Expansion Phase: TAK-580 NRAS WT+ Naive
Started | 4 | 3 | 3 | 3 | 7 | 7 | 3 | 3 | 13 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 4 | 3 | 3 | 3 | 7 | 7 | 3 | 3 | 13 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Progressive Disease | 2 | 3 | 2 | 3 | 5 | 4 | 0 | 2 | 6 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Unsatisfactory Therapeutic Response | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Symptomatic Deterioration | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Dose Expansion Phase
Arm/Group | Q2D Dose Escalation Phase: TAK-580 20 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 40 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 80 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 135 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 200 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 280 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 200 mg (28 Days Cycle) | QW Dose Escalation Phase: TAK-580 400 mg (28 Days Cycle) | QW Dose Escalation Phase: TAK-580 600 mg (28 Days Cycle) | QW Dose Escalation Phase: TAK-580 800 mg (28 Days Cycle) | Q2D Dose Expansion Phase: TAK-580 (BRAF+ Naive) | Q2D Dose Expansion Phase: TAK-580 (BRAF+ Previously Treated) | Q2D Dose Expansion Phase: TAK-580 (NRAS+ Naive) | Q2D Dose Expansion Phase: TAK-580 (NRAS+ Previously Treated) | Q2D Dose Expansion Phase: TAK-580 BRAF/NRAS WT+ Naive | Q2D Dose Expansion Phase:TAK-580 BRAF/NRASWT+PreviouslyTreated | Q2D Dose Expansion Phase: Pharmacokinetic Cohort | Q2D Dose Expansion Phase: TAK-580 (BRAF+) | QW Dose Expansion Phase: TAK-580 NRAS WT+ Naive
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16 | 8 | 16 | 1 | 6 | 11 | 20 | 2 | 19
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 15 | 8 | 16 | 1 | 6 | 11 | 20 | 2 | 19
Not completed — Progressive Disease | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 4 | 12 | 1 | 5 | 8 | 9 | 2 | 10
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 4
Not completed — Symptomatic Deterioration | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 3 | 0 | 1 | 1 | 5 | 0 | 3
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Unsatisfactory Therapeutic Response | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least 1 dose of study drug (TAK-580).
Groups:
- Q2D Dose Escalation Phase: TAK-580 20 mg (22 Days Cycle): TAK-580 20 mg, tablet, orally, Q2D, in each 22-days treatment cycle until disease progression, unacceptable toxicity, or participant discontinuation for any other reason (up to Cycle 38).
- Q2D Dose Escalation Phase: TAK-580 40 mg (22 Days Cycle): TAK-580 40 mg, tablet, orally, Q2D, in each 22-days treatment cycle until disease progression, unacceptable toxicity, or participant discontinuation for any other reason (up to Cycle 38).
- Q2D Dose Escalation Phase: TAK-580 80 mg (22 Days Cycle): TAK-580 80 mg, tablet, orally, Q2D, in each 22-days treatment cycle until disease progression, unacceptable toxicity, or participant discontinuation for any other reason (up to Cycle 38).
- Q2D Dose Expansion Phase: TAK-580 (BRAF+ Naive): TAK-580 200 mg, tablets, orally, Q2D, in each 28-days treatment cycle until disease progression, unacceptable toxicity, or participant discontinuation for any other reason (up to Cycle 49) in participants with BRAF mutation-positive cutaneous melanoma, naive to prior therapy with RAF and MEK inhibitors.
- Q2D Dose Expansion Phase: TAK-580 BRAF/NRAS WT+ Naive: TAK-580 200 mg, tablets, orally, Q2D, in each 28-days treatment cycle until disease progression, unacceptable toxicity, or participant discontinuation for any other reason (up to Cycle 49) in participants with BRAF/NRAS mutation-negative cutaneous melanoma (WT), naive to any prior anticancer therapy except ipilimumab, PD-1, and PDL-1 monoclonal antibodies.
- Total: Total of all reporting groups
Arm/Group | Q2D Dose Escalation Phase: TAK-580 20 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 40 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 80 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 135 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 200 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 280 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 200 mg (28 Days Cycle) | QW Dose Escalation Phase: TAK-580 400 mg (28 Days Cycle) | QW Dose Escalation Phase: TAK-580 600 mg (28 Days Cycle) | QW Dose Escalation Phase: TAK-580 800 mg (28 Days Cycle) | Q2D Dose Expansion Phase: TAK-580 (BRAF+ Naive) | Q2D Dose Expansion Phase: TAK-580 (BRAF+ Previously Treated) | Q2D Dose Expansion Phase: TAK-580 (NRAS+ Naive) | Q2D Dose Expansion Phase: TAK-580 (NRAS+ Previously Treated) | Q2D Dose Expansion Phase: TAK-580 BRAF/NRAS WT+ Naive | Q2D Dose Expansion Phase:TAK-580 BRAF/NRASWT+PreviouslyTreated | Q2D Dose Expansion Phase: Pharmacokinetic Cohort | Q2D Dose Expansion Phase: TAK-580 (BRAF+) | QW Dose Expansion Phase: TAK-580 NRAS WT+ Naive | Total
Number analyzed (Participants) | 4 | 3 | 3 | 3 | 7 | 7 | 3 | 3 | 13 | 4 | 16 | 8 | 16 | 1 | 6 | 11 | 20 | 2 | 19 | 149
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.0 (10.10) | 66.3 (8.33) | 56.7 (10.26) | 54.7 (13.65) | 58.7 (14.77) | 65.0 (4.40) | 71.0 (6.24) | 54.7 (13.58) | 57.2 (9.34) | 66.8 (7.50) | 54.6 (12.44) | 58.9 (16.39) | 68.4 (7.86) | 56.0 (NA) — Standard deviation could not be calculated because only one participant was analysed. | 56.7 (17.24) | 67.5 (8.69) | 65.1 (14.67) | 50.5 (0.71) | 66.1 (11.13) | 62.5 (12.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 2 | 2 | 1 | 4 | 2 | 1 | 8 | 2 | 6 | 5 | 6 | 1 | 3 | 6 | 8 | 2 | 9 | 73
  Male | 1 | 1 | 1 | 1 | 6 | 3 | 1 | 2 | 5 | 2 | 10 | 3 | 10 | 0 | 3 | 5 | 12 | 0 | 10 | 76
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 1 | 0 | 1 | 2 | 0 | 2 | 4 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 16
  Not Hispanic or Latino | 1 | 1 | 1 | 1 | 3 | 2 | 3 | 1 | 9 | 3 | 14 | 7 | 16 | 1 | 6 | 11 | 17 | 2 | 18 | 117
  Unknown or Not Reported | 1 | 1 | 1 | 2 | 3 | 3 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5
  White | 3 | 3 | 3 | 2 | 6 | 6 | 3 | 3 | 12 | 3 | 15 | 8 | 16 | 1 | 6 | 11 | 19 | 2 | 19 | 141
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 3 | 3 | 3 | 7 | 7 | 3 | 3 | 13 | 4 | 6 | 0 | 10 | 0 | 1 | 4 | 20 | 0 | 11 | 102
  United Kingdom | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 8 | 6 | 1 | 5 | 7 | 0 | 2 | 8 | 47

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting One or More Treatment-emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs) and Deaths
Time Frame: Baseline up to 30 days after last dose, or start of subsequent therapy, whichever occurred first (up to Cycle 38 Days 52 [Q2D] and 58 [QW] [Cycle=22 days (Q2D) and 28 days (QW)] in Escalation Phase; Cycle 49 Day 58 [Cycle=28 days] in Expansion Phase)
Population: The safety population included all participants who received at least 1 dose of study drug (TAK-580).
Measure: Count of Participants; unit: Participants
Arm/Group | Q2D Dose Escalation Phase: TAK-580 20 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 40 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 80 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 135 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 200 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 280 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 200 mg (28 Days Cycle) | QW Dose Escalation Phase: TAK-580 400 mg (28 Days Cycle) | QW Dose Escalation Phase: TAK-580 600 mg (28 Days Cycle) | QW Dose Escalation Phase: TAK-580 800 mg (28 Days Cycle) | Q2D Dose Expansion Phase: TAK-580 (BRAF+ Naive) | Q2D Dose Expansion Phase: TAK-580 (BRAF+ Previously Treated) | Q2D Dose Expansion Phase: TAK-580 (NRAS+ Naive) | Q2D Dose Expansion Phase: TAK-580 (NRAS+ Previously Treated) | Q2D Dose Expansion Phase: TAK-580 BRAF/NRAS WT+ Naive | Q2D Dose Expansion Phase:TAK-580 BRAF/NRASWT+PreviouslyTreated | Q2D Dose Expansion Phase: Pharmacokinetic Cohort | QW Dose Expansion Phase: TAK-580 NRAS WT+ Naive | Q2D Dose Expansion Phase: TAK-580 (BRAF+)
Number analyzed (Participants) | 4 | 3 | 3 | 3 | 7 | 7 | 3 | 3 | 13 | 4 | 16 | 8 | 16 | 1 | 6 | 11 | 20 | 19 | 2
Participants
  TEAEs | 4 | 3 | 3 | 3 | 7 | 7 | 3 | 3 | 13 | 4 | 16 | 8 | 16 | 1 | 6 | 11 | 20 | 19 | 2
  SAEs | 2 | 0 | 1 | 0 | 2 | 4 | 1 | 2 | 5 | 3 | 9 | 6 | 5 | 1 | 2 | 4 | 11 | 8 | 2
  Deaths | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 2 | 2 | 0 | 0 | 0 | 1 | 0 | 1

2. Primary Outcome: Dose Escalation Phase: Number of Participants With Dose-limiting Adverse Events (AEs)
Description: Dose limiting AEs were evaluated according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.03. Dose limiting AEs were defined as any of the following events: Grade 4 neutropenia for more than 7 days under maximum supportive therapy; febrile neutropenia; platelet counts decreased of Grade 3 requiring platelet transfusion or blood platelet decreased of Grade 4; if Course 2 was not initiated within 14 days due to AE related to the protocol treatment; Grade 3 or higher non-hematologic toxicity that was considered clinically significant, except the following cases, Grade 3 gastrointestinal symptoms that could be controlled with supportive therapy (example, appropriate use of antiemetics, antidiarrheals), and Grade 3 or higher electrolyte abnormalities that were not deemed clinically significant.
Time Frame: Cycle 1 (Cycle length= 22 days [Q2D] and 28 days [QW])
Population: The safety population included all participants who received at least 1 dose of study drug (TAK-580).
Measure: Count of Participants; unit: Participants
Arm/Group | Q2D Dose Escalation Phase: TAK-580 20 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 40 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 80 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 135 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 200 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 280 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 200 mg (28 Days Cycle) | QW Dose Escalation Phase: TAK-580 400 mg (28 Days Cycle) | QW Dose Escalation Phase: TAK-580 600 mg (28 Days Cycle) | QW Dose Escalation Phase: TAK-580 800 mg (28 Days Cycle)
Number analyzed (Participants) | 4 | 3 | 3 | 3 | 7 | 7 | 3 | 3 | 13 | 4
Participants | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2

3. Primary Outcome: Number of Participants With TEAEs Related to Physical Examination Findings
Time Frame: as for outcome 1
Population: The safety population included all participants who received at least 1 dose of study drug (TAK-580).
Measure: Count of Participants; unit: Participants
Arm/Group | Q2D Dose Escalation Phase: TAK-580 20 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 40 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 80 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 135 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 200 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 280 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 200 mg (28 Days Cycle) | QW Dose Escalation Phase: TAK-580 400 mg (28 Days Cycle) | QW Dose Escalation Phase: TAK-580 600 mg (28 Days Cycle) | QW Dose Escalation Phase: TAK-580 800 mg (28 Days Cycle) | Q2D Dose Expansion Phase: TAK-580 (BRAF+ Naive) | Q2D Dose Expansion Phase: TAK-580 (BRAF+ Previously Treated) | Q2D Dose Expansion Phase: TAK-580 (NRAS+ Naive) | Q2D Dose Expansion Phase: TAK-580 (NRAS+ Previously Treated) | Q2D Dose Expansion Phase: TAK-580 BRAF/NRAS WT+ Naive | Q2D Dose Expansion Phase:TAK-580 BRAF/NRASWT+PreviouslyTreated | Q2D Dose Expansion Phase: Pharmacokinetic Cohort | QW Dose Expansion Phase: TAK-580 NRAS WT+ Naive | Q2D Dose Expansion Phase: TAK-580 (BRAF+)
Number analyzed (Participants) | 4 | 3 | 3 | 3 | 7 | 7 | 3 | 3 | 13 | 4 | 16 | 8 | 16 | 1 | 6 | 11 | 20 | 19 | 2
Participants
  Weight decreased | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 1 | 2 | 1 | 2 | 0
  Weight increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 0
  Breath sounds abnormal | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Clinically Significant Change From Baseline in Body Weight at End of Study Visit (EOSV)
Time Frame: Baseline up to EOSV (up to Cycle 38 Days 52 [Q2D] and 58 [QW] [Cycle length =22 days (Q2D) and 28 days (QW)] in Escalation Phase; Cycle 49 Day 58 [Cycle length =28 days] in Expansion Phase)
Population: The safety population included all participants who received at least 1 dose of study drug (TAK-580). Participants who were evaluable for this measure at given time point were included for the assessment.
Measure: Mean (Standard Deviation); unit: kilogram (kg)
Arm/Group | Q2D Dose Escalation Phase: TAK-580 20 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 40 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 80 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 135 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 200 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 280 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 200 mg (28 Days Cycle) | QW Dose Escalation Phase: TAK-580 400 mg (28 Days Cycle) | QW Dose Escalation Phase: TAK-580 600 mg (28 Days Cycle) | QW Dose Escalation Phase: TAK-580 800 mg (28 Days Cycle) | Q2D Dose Expansion Phase: TAK-580 (BRAF+ Naive) | Q2D Dose Expansion Phase: TAK-580 (BRAF+ Previously Treated) | Q2D Dose Expansion Phase: TAK-580 (NRAS+ Naive) | Q2D Dose Expansion Phase: TAK-580 (NRAS+ Previously Treated) | Q2D Dose Expansion Phase: TAK-580 BRAF/NRAS WT+ Naive | Q2D Dose Expansion Phase:TAK-580 BRAF/NRASWT+PreviouslyTreated | Q2D Dose Expansion Phase: Pharmacokinetic Cohort | QW Dose Expansion Phase: TAK-580 NRAS WT+ Naive | Q2D Dose Expansion Phase: TAK-580 (BRAF+)
Number analyzed (Participants) | 4 | 3 | 3 | 3 | 7 | 7 | 3 | 3 | 13 | 4 | 16 | 8 | 16 | 1 | 6 | 11 | 20 | 19 | 2
kilogram (kg)
  Baseline: number analyzed (Participants) | 4 | 3 | 3 | 3 | 7 | 7 | 3 | 3 | 13 | 4 | 16 | 8 | 16 | 1 | 6 | 11 | 20 | 19 | 1
  Baseline | 87.477 (15.7794) | 72.077 (8.2162) | 67.375 (17.3371) | 77.717 (4.1695) | 76.963 (21.9026) | 77.695 (14.3247) | 69.522 (17.6937) | 73.589 (13.2534) | 81.054 (23.6907) | 80.503 (15.7401) | 95.837 (30.2887) | 71.288 (8.6570) | 81.312 (17.4736) | 57.100 (NA) — Standard deviation could not be calculated because only one participant was evaluable | 75.267 (15.3231) | 72.847 (23.8439) | 79.624 (16.6098) | 83.298 (16.3695) | 67.000 (NA) — Standard deviation could not be calculated because only one participant was evaluable
  Change at EOSV: number analyzed (Participants) | 3 | 3 | 3 | 3 | 7 | 4 | 2 | 3 | 10 | 2 | 13 | 3 | 9 | 0 | 6 | 7 | 14 | 16 | 0
  Change at EOSV | 7.167 (16.0315) | -1.693 (1.4468) | 1.542 (1.1139) | -0.907 (1.3698) | 0.065 (1.4543) | -0.544 (3.1033) | 0.272 (1.6037) | -1.225 (4.5746) | -1.868 (4.8255) | -1.270 (0.0005) | -7.825 (20.1782) | -1.700 (6.2386) | -3.164 (3.7607) |  | -3.225 (2.9826) | 0.201 (3.7358) | -4.292 (6.5671) | -3.189 (3.9690) |

5. Primary Outcome: Number of Participants With Abnormal Clinically Significant Electrocardiogram (ECG) Findings
Time Frame: as for outcome 1
Population: The safety population included all participants who received at least 1 dose of study drug (TAK-580).
Measure: Count of Participants; unit: Participants
Arm/Group | Q2D Dose Escalation Phase: TAK-580 20 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 40 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 80 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 135 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 200 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 280 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 200 mg (28 Days Cycle) | QW Dose Escalation Phase: TAK-580 400 mg (28 Days Cycle) | QW Dose Escalation Phase: TAK-580 600 mg (28 Days Cycle) | QW Dose Escalation Phase: TAK-580 800 mg (28 Days Cycle) | Q2D Dose Expansion Phase: TAK-580 (BRAF+ Naive) | Q2D Dose Expansion Phase: TAK-580 (BRAF+ Previously Treated) | Q2D Dose Expansion Phase: TAK-580 (NRAS+ Naive) | Q2D Dose Expansion Phase: TAK-580 (NRAS+ Previously Treated) | Q2D Dose Expansion Phase: TAK-580 BRAF/NRAS WT+ Naive | Q2D Dose Expansion Phase:TAK-580 BRAF/NRASWT+PreviouslyTreated | Q2D Dose Expansion Phase: Pharmacokinetic Cohort | QW Dose Expansion Phase: TAK-580 NRAS WT+ Naive | Q2D Dose Expansion Phase: TAK-580 (BRAF+)
Number analyzed (Participants) | 4 | 3 | 3 | 3 | 7 | 7 | 3 | 3 | 13 | 4 | 16 | 8 | 16 | 1 | 6 | 11 | 20 | 19 | 2
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Eastern Cooperative Oncology Group (ECOG) Performance Score
Description: ECOG performance score was measured on 6 point scale to assess participant's performance status, where: 0 (fully active, able to carry on all pre-disease activities without restriction); 1 (restricted in physically strenuous activity, but ambulatory and able to carry out light or sedentary work); 2 (ambulatory greater than(>) 50 percent (%) of waking hours), capable of all self-care, unable to carry out any work activities); 3 (capable of only limited self-care, confined to bed or chair >50% of waking hours); 4(completely disabled, cannot carry on any self-care, totally confined to bed or chair); 5 (dead). A higher score indicated greater functional impairment.
Time Frame: at EOSV (up to Cycle 38 Days 52 [Q2D] and 58 [QW] [Cycle length =22 days (Q2D) and 28 days (QW)] in Escalation Phase; Cycle 49 Day 58 [Cycle length =28 days] in Expansion Phase)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Q2D Dose Escalation Phase: TAK-580 20 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 40 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 80 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 135 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 200 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 280 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 200 mg (28 Days Cycle) | QW Dose Escalation Phase: TAK-580 400 mg (28 Days Cycle) | QW Dose Escalation Phase: TAK-580 600 mg (28 Days Cycle) | QW Dose Escalation Phase: TAK-580 800 mg (28 Days Cycle) | Q2D Dose Expansion Phase: TAK-580 (BRAF+ Naive) | Q2D Dose Expansion Phase: TAK-580 (BRAF+ Previously Treated) | Q2D Dose Expansion Phase: TAK-580 (NRAS+ Naive) | Q2D Dose Expansion Phase: TAK-580 (NRAS+ Previously Treated) | Q2D Dose Expansion Phase: TAK-580 BRAF/NRAS WT+ Naive | Q2D Dose Expansion Phase:TAK-580 BRAF/NRASWT+PreviouslyTreated | Q2D Dose Expansion Phase: Pharmacokinetic Cohort | QW Dose Expansion Phase: TAK-580 NRAS WT+ Naive | Q2D Dose Expansion Phase: TAK-580 (BRAF+)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 7 | 5 | 2 | 3 | 10 | 2 | 14 | 4 | 12 | 0 | 6 | 11 | 14 | 15 | 1
score on a scale | 1.0 (0.00) | 1.0 (1.00) | 1.7 (1.53) | 0.3 (0.58) | 1.3 (0.49) | 1.2 (0.45) | 1.0 (0.00) | 0.7 (0.58) | 1.0 (0.47) | 1.0 (0.00) | 0.7 (0.73) | 1.5 (0.58) | 0.6 (0.90) |  | 0.8 (0.41) | 1.2 (0.98) | 0.6 (0.74) | 0.7 (0.80) | 2.0 (NA) — Standard deviation could not be calculated because only one participant was evaluable

7. Primary Outcome: Number of Participants With TEAEs Categorized Into Investigations Related to Laboratory Test of Chemistry, Hematology or Urinalysis
Time Frame: as for outcome 1
Population: The safety population included all participants who received at least 1 dose of study drug (TAK-580).
Measure: Count of Participants; unit: Participants
Arm/Group | Q2D Dose Escalation Phase: TAK-580 20 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 40 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 80 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 135 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 200 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 280 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 200 mg (28 Days Cycle) | QW Dose Escalation Phase: TAK-580 400 mg (28 Days Cycle) | QW Dose Escalation Phase: TAK-580 600 mg (28 Days Cycle) | QW Dose Escalation Phase: TAK-580 800 mg (28 Days Cycle) | Q2D Dose Expansion Phase: TAK-580 (BRAF+ Naive) | Q2D Dose Expansion Phase: TAK-580 (BRAF+ Previously Treated) | Q2D Dose Expansion Phase: TAK-580 (NRAS+ Naive) | Q2D Dose Expansion Phase: TAK-580 (NRAS+ Previously Treated) | Q2D Dose Expansion Phase: TAK-580 BRAF/NRAS WT+ Naive | Q2D Dose Expansion Phase:TAK-580 BRAF/NRASWT+PreviouslyTreated | Q2D Dose Expansion Phase: Pharmacokinetic Cohort | QW Dose Expansion Phase: TAK-580 NRAS WT+ Naive | Q2D Dose Expansion Phase: TAK-580 (BRAF+)
Number analyzed (Participants) | 4 | 3 | 3 | 3 | 7 | 7 | 3 | 3 | 13 | 4 | 16 | 8 | 16 | 1 | 6 | 11 | 20 | 19 | 2
Participants
  Liver function analyses | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 5 | 0 | 3 | 3 | 5 | 2 | 2
  Skeletal and cardiac muscle analyses | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 1 | 2 | 0 | 0 | 5 | 6 | 1 | 1
  Mineral and electrolyte analyses | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 0 | 0 | 0 | 0 | 2 | 1 | 1
  Tissue enzyme analyses NEC | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 2 | 1 | 0 | 1
  Renal function analyses | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 4 | 0 | 0
  Platelet analyses | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 0
  White blood cell analyses | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1
  Red blood cell analyses | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Pituitary analyses anterior | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Carbohydrate tolerance analyses (incl diabetes) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Cardiac function diagnostic procedures | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Coagulation and bleeding analyses | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Digestive enzymes | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR was defined as the percentage of participants with complete response (CR) or partial response (PR). The ORR assessment was based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. CR: was disappearance of all target lesions. Any pathological lymph nodes (target or non-target) had to be reduced in short axis to less than (<) 10 millimeter (mm). PR: was at least a 30% decrease in sum of diameter (SOD) of target lesions, taking as reference the baseline SOD.
Time Frame: as for outcome 4
Population: Response-evaluable population included all participants with measurable disease who received any amount of TAK-580 and had at least 1 postbaseline response assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Q2D Dose Escalation Phase: TAK-580 20 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 40 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 80 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 135 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 200 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 280 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 200 mg (28 Days Cycle) | QW Dose Escalation Phase: TAK-580 400 mg (28 Days Cycle) | QW Dose Escalation Phase: TAK-580 600 mg (28 Days Cycle) | QW Dose Escalation Phase: TAK-580 800 mg (28 Days Cycle) | Q2D Dose Expansion Phase: TAK-580 (BRAF+ Naive) | Q2D Dose Expansion Phase: TAK-580 (BRAF+ Previously Treated) | Q2D Dose Expansion Phase: TAK-580 (NRAS+ Naive) | Q2D Dose Expansion Phase: TAK-580 (NRAS+ Previously Treated) | Q2D Dose Expansion Phase: TAK-580 BRAF/NRAS WT+ Naive | Q2D Dose Expansion Phase:TAK-580 BRAF/NRASWT+PreviouslyTreated | Q2D Dose Expansion Phase: Pharmacokinetic Cohort | QW Dose Expansion Phase: TAK-580 NRAS WT+ Naive | Q2D Dose Expansion Phase: TAK-580 (BRAF+)
Number analyzed (Participants) | 3 | 3 | 2 | 3 | 6 | 4 | 1 | 3 | 8 | 3 | 16 | 6 | 14 | 1 | 6 | 9 | 14 | 17 | 2
percentage of participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 13 | 33 | 50 | 17 | 7 | 0 | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was the time from first dose date of study drug to date of the first documentation of confirmed progressive disease (PD) or death, whichever occurred first. The PFS assessment was based on RECIST 1.1. PD: at least 20% increase (including an absolute increase of at least 5 mm) in the SOD of target lesions. PFS was calculated using Kaplan-Meier estimate and presented with 2-sided 95% confidence interval. Participants with no response assessment were censored at the date of first dose.
Time Frame: Baseline up to the date of first document PD, or death due to any cause, whichever occurred first (up to Cycle 38 Days 52 [Q2D] and 58 [QW] [Cycle =22 days (Q2D) and 28 days (QW)] in Escalation Phase; Cycle 49 Day 58 [Cycle =28 days] in Expansion Phase)
Population: The safety population included all participants who received at least 1 dose of study drug (TAK-580).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Q2D Dose Escalation Phase: TAK-580 20 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 40 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 80 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 135 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 200 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 280 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 200 mg (28 Days Cycle) | QW Dose Escalation Phase: TAK-580 400 mg (28 Days Cycle) | QW Dose Escalation Phase: TAK-580 600 mg (28 Days Cycle) | QW Dose Escalation Phase: TAK-580 800 mg (28 Days Cycle) | Q2D Dose Expansion Phase: TAK-580 (BRAF+ Naive) | Q2D Dose Expansion Phase: TAK-580 (BRAF+ Previously Treated) | Q2D Dose Expansion Phase: TAK-580 (NRAS+ Naive) | Q2D Dose Expansion Phase: TAK-580 (NRAS+ Previously Treated) | Q2D Dose Expansion Phase: TAK-580 BRAF/NRAS WT+ Naive | Q2D Dose Expansion Phase:TAK-580 BRAF/NRASWT+PreviouslyTreated | Q2D Dose Expansion Phase: Pharmacokinetic Cohort | QW Dose Expansion Phase: TAK-580 NRAS WT+ Naive | Q2D Dose Expansion Phase: TAK-580 (BRAF+)
Number analyzed (Participants) | 4 | 3 | 3 | 3 | 7 | 7 | 3 | 3 | 13 | 4 | 16 | 8 | 16 | 1 | 6 | 11 | 20 | 19 | 2
months | 1.4 [0.8 to NA] — Upper limit of confidence interval could not be calculated because 75% of the participants had an event. | 1.4 [1.0 to 1.4] | 1.4 [1.0 to 1.5] | 1.4 [1.4 to 1.4] | 1.5 [1.3 to 2.8] | 1.2 [0.9 to 32.5] | NA [NA to NA] — Median, lower and upper limit of confidence interval could not be calculated because no participant had an event | 9.2 [0.8 to 9.2] | 1.5 [0.7 to 1.9] | 1.9 [1.0 to NA] — Upper limit of confidence interval could not be calculated because 75% of the participants had an event. | 5.7 [1.9 to 14.3] | 2.4 [1.0 to 3.7] | 1.8 [1.8 to 3.2] | 0.8 [NA to NA] — Confidence interval could not be calculated due to low number of events. | 1.9 [1.8 to 2.2] | 1.8 [1.7 to 5.5] | 3.6 [1.8 to NA] — Upper limit of confidence interval could not be calculated because 50% of the participants were censored. | 2.3 [1.9 to 5.5] | 1.7 [1.6 to 1.8]

10. Secondary Outcome: Duration of Response (DOR)
Description: DOR was assessed from the first documented response (CR or PR) to the date of first documented PD and was censored at the date of the last assessment for responders who died without documented PD and for responders who were still alive and had not progressed. DOR assessment was based on RECIST v1.1. CR: was disappearance of all target lesions. Any pathological lymph nodes (target or non-target) had to be reduced in short axis to <10 mm. PR: at least 30% decrease in SOD of target lesions, taking as reference the baseline SOD persistence of one or more non-target lesions and/or maintenance of tumor marker level above the normal limits. PD: at least 20% increase (including an absolute increase of at least 5 mm) in the SOD of target lesions, taking as reference the smallest sum and/or unequivocal progression of existing non-target lesions and/or appearance of 1 or more new lesions. DOR was calculated using Kaplan-Meier estimate.
Time Frame: From the first documented response (CR or PR) up to the date of first documented PD (up to Cycle 38 Days 52 [Q2D] and 58 [QW] [Cycle =22 days (Q2D) and 28 days (QW)] in Escalation Phase; Cycle 49 Day 58 [Cycle =28 days] in Expansion Phase)
Population: Analysis population included only a subset of participants (all responders) with response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Q2D Dose Escalation Phase: TAK-580 20 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 40 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 80 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 135 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 200 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 280 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 200 mg (28 Days Cycle) | QW Dose Escalation Phase: TAK-580 400 mg (28 Days Cycle) | QW Dose Escalation Phase: TAK-580 600 mg (28 Days Cycle) | QW Dose Escalation Phase: TAK-580 800 mg (28 Days Cycle) | Q2D Dose Expansion Phase: TAK-580 (BRAF+ Naive) | Q2D Dose Expansion Phase: TAK-580 (BRAF+ Previously Treated) | Q2D Dose Expansion Phase: TAK-580 (NRAS+ Naive) | Q2D Dose Expansion Phase: TAK-580 (NRAS+ Previously Treated) | Q2D Dose Expansion Phase: TAK-580 BRAF/NRAS WT+ Naive | Q2D Dose Expansion Phase:TAK-580 BRAF/NRASWT+PreviouslyTreated | Q2D Dose Expansion Phase: Pharmacokinetic Cohort | QW Dose Expansion Phase: TAK-580 NRAS WT+ Naive | Q2D Dose Expansion Phase: TAK-580 (BRAF+)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 8 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
months |  |  |  |  |  |  |  |  | NA [NA to NA] — Median, lower and upper limit of confidence interval could not be calculated because no participant had an event | NA [NA to NA] — Median, lower and upper limit of confidence interval could not be calculated because no participant had an event | 6.0 [3.7 to NA] — Upper limit of confidence interval could not be calculated because 63% of the participants had an event | NA [NA to NA] — Median, lower and upper limit of confidence interval could not be calculated because no participant had an event | 1.5 [NA to NA] — Confidence interval could not be calculated due to low number of events. |  |  |  |  |  |

11. Secondary Outcome: Dose Escalation Phase and Dose Expansion Pharmacokinetic Cohort, Cmax: Maximum Observed Plasma Concentration for TAK-580
Time Frame: Escalation (Esc.) and Expansion (Exp.) Q2D: C1D1 and 21 pre-dose and at multiple time points (up to 48 hours [h]) post-dose (C=22 days [Esc. Q2D] and 28 days [Exp. Q2D]); Esc. QW: C1D1 and 22 at multiple time-points (up to168 h) post-dose (C=28 days)
Population: The PK-evaluable population included all participants who had sufficient dosing data and TAK-580 concentration-time data to permit calculation of any TAK-580 parameters. PK-evaluable population where data at specified time points was available.
Measure: Geometric Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Q2D Dose Escalation Phase: TAK-580 20 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 40 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 80 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 135 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 200 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 280 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 200 mg (28 Days Cycle) | QW Dose Escalation Phase: TAK-580 400 mg (28 Days Cycle) | QW Dose Escalation Phase: TAK-580 600 mg (28 Days Cycle) | QW Dose Escalation Phase: TAK-580 800 mg (28 Days Cycle) | Q2D Dose Expansion Phase: Pharmacokinetic Cohort
Number analyzed (Participants) | 4 | 3 | 3 | 3 | 7 | 7 | 3 | 3 | 13 | 4 | 20
nanogram per milliliter (ng/mL)
  Cycle 1 Day 1 | 140.0 (86.61) | 393.1 (49.81) | 921.7 (332.40) | 1048.1 (290.91) | 1933.6 (717.03) | 2675.2 (1296.95) | 2072.8 (287.29) | 2934.0 (690.39) | 4459.3 (1475.08) | 6774.3 (1082.79) | 1606.9 (670.48)
  Cycle 1 Day 21: number analyzed (Participants) | 3 | 2 | 3 | 3 | 6 | 4 | 2 | 0 | 0 | 0 | 12
  Cycle 1 Day 21 | 301.5 (61.83) | 759.7 (138.59) | 2038.8 (1076.99) | 3321.5 (1275.83) | 3809.1 (466.85) | 4063.1 (782.33) | 4588.4 (700.04) |  |  |  | 3548.8 (1310.21)
  Cycle 1 Day 22: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 6 | 3 | 0
  Cycle 1 Day 22 |  |  |  |  |  |  |  | 3135.2 (485.70) | 4739.8 (2902.53) | 6460.2 (1632.31) |

12. Secondary Outcome: Dose Escalation Phase and Dose Expansion Pharmacokinetic Cohort, Ctrough: Trough Concentration for TAK-580
Time Frame: Escalation and Expansion Q2D Cohorts: C1D21 pre-dose (C=22 days [Escalation Q2D] and 28 days [Expansion Q2D]); Escalation QW Cohorts: C1D22 pre-dose (C= 28 days)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Q2D Dose Escalation Phase: TAK-580 20 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 40 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 80 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 135 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 200 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 280 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 200 mg (28 Days Cycle) | QW Dose Escalation Phase: TAK-580 400 mg (28 Days Cycle) | QW Dose Escalation Phase: TAK-580 600 mg (28 Days Cycle) | QW Dose Escalation Phase: TAK-580 800 mg (28 Days Cycle) | Q2D Dose Expansion Phase: Pharmacokinetic Cohort
Number analyzed (Participants) | 4 | 3 | 3 | 3 | 7 | 7 | 3 | 3 | 13 | 4 | 20
ng/mL
  Cycle 1 Day 21: number analyzed (Participants) | 3 | 2 | 3 | 3 | 6 | 4 | 2 | 0 | 0 | 0 | 12
  Cycle 1 Day 21 | 178.3 (42.92) | 265.5 (74.25) | 1080.0 (797.75) | 1720.0 (708.87) | 1739.7 (746.88) | 2135.0 (494.00) | 2700.0 (1088.94) |  |  |  | 2085.0 (672.26)
  Cycle 1 Day 22: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 6 | 3 | 0
  Cycle 1 Day 22 |  |  |  |  |  |  |  | 270.0 (108.00) | 898.7 (618.68) | 1216.7 (841.80) |

13. Secondary Outcome: Dose Escalation Phase and Dose Expansion Pharmacokinetic Cohort, Tmax: Time to Reach the Cmax for TAK-580
Time Frame: Escalation (Esc.) and Expansion (Exp.) Q2D: C1D1 and 21 pre-dose and at multiple time points (up to 48 h) post-dose (C=22 days [Esc. Q2D] and 28 days [Exp. Q2D]); Esc. QW: C1D1 and 22 at multiple time-points (up to168 h) post-dose (C=28 days)
Population: as for outcome 11
Measure: Median (Full Range); unit: hour
Arm/Group | Q2D Dose Escalation Phase: TAK-580 20 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 40 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 80 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 135 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 200 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 280 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 200 mg (28 Days Cycle) | QW Dose Escalation Phase: TAK-580 400 mg (28 Days Cycle) | QW Dose Escalation Phase: TAK-580 600 mg (28 Days Cycle) | QW Dose Escalation Phase: TAK-580 800 mg (28 Days Cycle) | Q2D Dose Expansion Phase: Pharmacokinetic Cohort
Number analyzed (Participants) | 4 | 3 | 3 | 3 | 7 | 7 | 3 | 3 | 13 | 4 | 20
hour
  Cycle 1 Day 1: number analyzed (Participants) | 3 | 2 | 3 | 3 | 6 | 4 | 2 | 3 | 13 | 4 | 12
  Cycle 1 Day 1 | 3.983 [2.00 to 4.07] | 2.150 [1.98 to 4.05] | 2.033 [2.00 to 4.00] | 3.917 [1.18 to 4.02] | 2.050 [1.00 to 23.82] | 4.033 [0.97 to 23.00] | 4.000 [1.98 to 6.02] | 4.150 [3.20 to 5.12] | 3.150 [1.00 to 7.88] | 3.100 [2.12 to 7.27] | 3.108 [0.98 to 7.58]
  Cycle 1 Day 21: number analyzed (Participants) | 3 | 2 | 3 | 3 | 6 | 4 | 2 | 0 | 0 | 0 | 20
  Cycle 1 Day 21 | 2.000 [2.00 to 4.00] | 3.050 [2.10 to 4.00] | 4.050 [2.00 to 6.12] | 2.000 [1.00 to 2.00] | 2.992 [1.00 to 8.00] | 2.808 [1.98 to 4.00] | 12.792 [2.13 to 23.45] |  |  |  | 2.192 [1.87 to 6.17]
  Cycle 1 Day 22: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 6 | 3 | 0
  Cycle 1 Day 22 |  |  |  |  |  |  |  | 3.150 [2.80 to 3.17] | 3.033 [2.10 to 23.80] | 3.950 [2.87 to 7.32] |

14. Secondary Outcome: Dose Escalation Phase and Dose Expansion Pharmacokinetic Cohort, t1/2z: Terminal Phase Disposition Half-life for TAK-580
Time Frame: Escalation (Esc.) and Expansion (Exp.) Q2D: C1D21 pre-dose and at multiple time points (up to 48 h) post-dose (C=22 days [Esc. Q2D] and 28 days [Exp. Q2D]); Esc. QW: C1D22 at multiple time-points (up to168 h) post-dose (C=28 days)
Population: PK-evaluable population. t1/2z of TAK-580 could not be determined in cancer participants who were on Q2D regimen with a 48-hour dose interval since the duration of plasma PK sample collection within the dose interval was shorter than the anticipated t1/2z of TAK-580. PK-evaluable population where data at specified time points was available.
Measure: Median (Full Range); unit: hour
Arm/Group | Q2D Dose Escalation Phase: TAK-580 20 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 40 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 80 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 135 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 200 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 280 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 200 mg (28 Days Cycle) | QW Dose Escalation Phase: TAK-580 400 mg (28 Days Cycle) | QW Dose Escalation Phase: TAK-580 600 mg (28 Days Cycle) | QW Dose Escalation Phase: TAK-580 800 mg (28 Days Cycle) | Q2D Dose Expansion Phase: Pharmacokinetic Cohort
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 6 | 3 | 0
hour
  Cycle 1 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 1 Day 21: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 1 Day 22 |  |  |  |  |  |  |  | 50.22 [46.4 to 59.3] | 59.06 [31.1 to 119.2] | 69.65 [61.6 to 73.0] |

15. Secondary Outcome: Dose Escalation Phase and Dose Expansion Pharmacokinetic Cohort, CLr: Renal Clearance for TAK-580
Time Frame: Q2D Cohorts: Cycle1 Days 1 and 21 up to 24 hours post-dose (Cycle1 length= 22 days); QW Cohorts: Cycle2 Days 1 and 22 up to 7 hours post-dose (Cycle 2 length= 28 days)
Population: CLr of TAK-580 could not be determined since urine samples were collected for a limited duration during a site visit.
Arm/Group | Q2D Dose Escalation Phase: TAK-580 20 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 40 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 80 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 135 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 200 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 280 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 200 mg (28 Days Cycle) | QW Dose Escalation Phase: TAK-580 400 mg (28 Days Cycle) | QW Dose Escalation Phase: TAK-580 600 mg (28 Days Cycle) | QW Dose Escalation Phase: TAK-580 800 mg (28 Days Cycle) | Q2D Dose Expansion Phase: Pharmacokinetic Cohort
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

16. Secondary Outcome: Q2D Dose Escalation Phase and Q2D Dose Expansion Pharmacokinetic Cohort, AUC(0-48): Area Under the Plasma Concentration-time Curve From Time 0 to 48 Hours Postdose for TAK-580
Time Frame: Cycle 1 Days 1 and 21 pre-dose and at multiple time points (up to 48 hours) post-dose (Cycle length= 22 days)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | Q2D Dose Escalation Phase: TAK-580 20 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 40 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 80 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 135 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 200 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 280 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 200 mg (28 Days Cycle) | Q2D Dose Expansion Phase: Pharmacokinetic Cohort
Number analyzed (Participants) | 4 | 3 | 3 | 3 | 7 | 7 | 3 | 20
hour*nanogram per milliliter (h*ng/mL)
  Day 1 | 4799.7 (2570.95) | 11019.7 (655.03) | 30562.8 (16909.20) | 36061.9 (8904.40) | 50946.5 (10597.12) | 78993.3 (23713.60) | 66799.2 (7656.58) | 53522.2 (17337.54)
  Day 21: number analyzed (Participants) | 3 | 2 | 2 | 3 | 5 | 3 | 2 | 12
  Day 21 | 10679.2 (2571.83) | 21007.9 (3501.86) | 43294.2 (10403.72) | 99626.7 (29090.62) | 125540.2 (46299.79) | 156439.3 (26263.33) | 165002.1 (19899.97) | 127026.4 (38244.03)

17. Secondary Outcome: QW Dose Escalation Phase, AUC(0-168): Area Under the Plasma Concentration-time Curve From Time 0 to 168 Hours Postdose for TAK-580
Time Frame: Cycle 1 Days 1 and 22 pre-dose and at multiple time points (up to 168 hours) post-dose (Cycle length= 28 days)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | QW Dose Escalation Phase: TAK-580 400 mg (28 Days Cycle) | QW Dose Escalation Phase: TAK-580 600 mg (28 Days Cycle) | QW Dose Escalation Phase: TAK-580 800 mg (28 Days Cycle)
Number analyzed (Participants) | 3 | 13 | 4
h*ng/mL
  Day 1: number analyzed (Participants) | 3 | 10 | 4
  Day 1 | 184534.4 (50225.97) | 278247.9 (128772.92) | 431723.3 (106266.40)
  Day 22: number analyzed (Participants) | 3 | 6 | 3
  Day 22 | 199210.4 (57957.62) | 339244.8 (149201.72) | 477700.2 (86620.19)

18. Secondary Outcome: Dose Expansion Phase, Melanoma Cohorts: Percent Change From Baseline in RAF Inhibition Biomarkers at Specified Time Points
Description: The extent of phosphorylated extracellular signal-regulated kinase (pERK) staining was assessed in the melanoma expansion cohorts. The level of staining was assessed by a pathologist (semi-H scores) and by quantified image analysis (quant H-scores). The H-score scale used to interpret data from the pathologist rating was as follows: 0 to 99 =low staining; 100 to 199= medium staining; 200 to 300 =high staining. The H-score scale used to interpret data from the quantified image analysis was as followed: 0 to 100 =low staining; 100 to 150= medium staining; 150 to 235= high staining.
Time Frame: Baseline, Cycle 1 Day 21 (Q2D), and Cycle 1 Day 22 (QW) (Cycle length= 22 days [Q2D] and 28 days [QW])
Population: Pharmacodynamic (PD)-evaluable: all participants who had sufficient dosing and PD data,collected within protocol-specified window of sampling time.Participants who were evaluable for this measure at given time point were included. Data for this measure was not planned to be collected and analyzed for Q2D Dose Expansion Phase:Pharmacokinetic Cohort.
Measure: Median (Full Range); unit: percent change
Arm/Group | Q2D Dose Expansion Phase: TAK-580 (BRAF+ Naive) | Q2D Dose Expansion Phase: TAK-580 (BRAF+ Previously Treated) | Q2D Dose Expansion Phase: TAK-580 (NRAS+ Naive) | Q2D Dose Expansion Phase: TAK-580 (NRAS+ Previously Treated) | Q2D Dose Expansion Phase: TAK-580 BRAF/NRAS WT+ Naive | Q2D Dose Expansion Phase:TAK-580 BRAF/NRASWT+PreviouslyTreated | QW Dose Expansion Phase: TAK-580 NRAS WT+ Naive | Q2D Dose Expansion Phase: TAK-580 (BRAF+)
Number analyzed (Participants) | 3 | 4 | 6 | 0 | 2 | 5 | 3 | 1
percent change
  Quant H-score: number analyzed (Participants) | 2 | 4 | 5 | 0 | 2 | 5 | 1 | 1
  Quant H-score | 180.0 [-100 to 460] | -93.5 [-97 to 1235] | -82.0 [-96 to -43] |  | -51.0 [-97 to -5] | -15.0 [-95 to 22] | -8.0 [-8 to -8] | -71.0 [-71 to -71]
  Semi H-score: number analyzed (Participants) | 2 | 4 | 5 | 0 | 2 | 5 | 1 | 1
  Semi H-score | -94.5 [-100 to -89] | -80.5 [-100 to 2207] | -70.0 [-100 to 603] |  | -24.5 [-78 to 29] | -27.0 [-100 to 0] | -12.0 [-12 to -12] | -23.0 [-23 to -23]

19. Secondary Outcome: Dose Expansion Phase, Melanoma Cohorts: Percent Change From Baseline in Apoptotic Biomarkers at Specified Time Points
Description: The extent of cleaved poly ADP-ribose polymerase (cPARP) and BIM-1 was assessed in the melanoma expansion cohorts. The level of staining was assessed by quantified image analysis (quant H-scores) and by quantified image analysis (quant H-scores). The H-score scale used to interpret data from the pathologist rating was as follows: 0 to 99= low staining; 100 to 199 =medium staining; 200 to 300 =high staining. The H-score scale used to interpret data from the quantified image analysis was as followed in cPARP: 0 to 70= low staining; 70 to 175 =medium staining; 175 to 240 =high staining; BIM-1: 0 to 128= low staining; 128 to 155 =medium staining; 155 to 229 =high staining.
Time Frame: Baseline, Cycle 1 Day 21 (Q2D), and Cycle 1 Day 22 (QW) (Cycle length= 22 days [Q2D] and 28 days [QW])
Population: PD-evaluable: all participants who had sufficient dosing and PD data, collected within protocol-specified window of sampling time. Participants who were evaluable for this measure at given time point were included. Data for this measure was not planned to be collected and analyzed for Q2D Dose Expansion Phase: Pharmacokinetic Cohort.
Measure: Median (Full Range); unit: percent change
Arm/Group | Q2D Dose Expansion Phase: TAK-580 (BRAF+ Naive) | Q2D Dose Expansion Phase: TAK-580 (BRAF+ Previously Treated) | Q2D Dose Expansion Phase: TAK-580 (NRAS+ Naive) | Q2D Dose Expansion Phase: TAK-580 (NRAS+ Previously Treated) | Q2D Dose Expansion Phase: TAK-580 BRAF/NRAS WT+ Naive | Q2D Dose Expansion Phase:TAK-580 BRAF/NRASWT+PreviouslyTreated | QW Dose Expansion Phase: TAK-580 NRAS WT+ Naive | Q2D Dose Expansion Phase: TAK-580 (BRAF+)
Number analyzed (Participants) | 3 | 4 | 6 | 0 | 2 | 5 | 3 | 1
percent change
  cPARP Quant H-score: number analyzed (Participants) | 0 | 4 | 3 | 0 | 1 | 4 | 0 | 0
  cPARP Quant H-score |  | -100.0 [-100 to -93] | 317.5 [-15 to 650] |  | -100.0 [-100 to -100] | -33.5 [-100 to 200] |  |
  cPARP Semi H-score: number analyzed (Participants) | 0 | 4 | 3 | 0 | 1 | 4 | 0 | 0
  cPARP Semi H-score |  | -96.0 [-100 to -92] | -33.0 [-33 to -33] |  | -11.0 [-11 to -11] | -48.0 [-100 to 0] |  |
  BIM-1 Quant H-score: number analyzed (Participants) | 3 | 4 | 4 | 0 | 2 | 4 | 2 | 1
  BIM-1 Quant H-score | 265.0 [265 to 265] | 136.0 [64 to 650] | 158.0 [90 to 625] |  | -52.5 [-65 to -40] | -23.5 [-53 to 66] | 35.5 [-29 to 100] | 960.0 [960 to 960]
  BIM-1 Semi H-score: number analyzed (Participants) | 1 | 4 | 4 | 0 | 2 | 4 | 2 | 0
  BIM-1 Semi H-score | 723.5 [47 to 1400] | 64.5 [-84 to 2533] | 64.0 [30 to 287] |  | -41.0 [-75 to -7] | -17.0 [-49 to 28] | -3.5 [-15 to 8] |

ADVERSE EVENTS:
Time Frame: TEAEs are AEs that started after the first dose of study drug and no more than 30 days after the last dose of study drug (approximately Cycle 38 Days 52 [Q2D] and 58 [QW] in Escalation Phase; Cycle 49 Day 58 in Expansion Phase)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Groups:
- Q2D Dose Escalation Phase: TAK-580 20 mg (22 Days Cycle): TAK-580 20 mg, tablets, orally, Q2D, in each 22-days treatment cycle until disease progression, unacceptable toxicity, or participant discontinuation for any other reason (up to Cy cle 38).
Arm/Group | Q2D Dose Escalation Phase: TAK-580 20 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 40 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 80 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 135 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 200 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 280 mg (22 Days Cycle) | Q2D Dose Escalation Phase: TAK-580 200 mg (28 Days Cycle) | QW Dose Escalation Phase: TAK-580 400 mg (28 Days Cycle) | QW Dose Escalation Phase: TAK-580 600 mg (28 Days Cycle) | QW Dose Escalation Phase: TAK-580 800 mg (28 Days Cycle) | Q2D Dose Expansion Phase: TAK-580 (BRAF+ Naive) | Q2D Dose Expansion Phase: TAK-580 (BRAF+ Previously Treated) | Q2D Dose Expansion Phase: TAK-580 (NRAS+ Naive) | Q2D Dose Expansion Phase: TAK-580 (NRAS+ Previously Treated) | Q2D Dose Expansion Phase: TAK-580 BRAF/NRAS WT+ Naive | Q2D Dose Expansion Phase:TAK-580 BRAF/NRASWT+PreviouslyTreated | Q2D Dose Expansion Phase: Pharmacokinetic Cohort | Q2D Dose Expansion Phase: TAK-580 (BRAF+) | QW Dose Expansion Phase: TAK-580 NRAS WT+ Naive
All-Cause Mortality (participants affected / at risk) | 1/4 | 0/3 | 1/3 | 0/3 | 0/7 | 1/7 | 0/3 | 0/3 | 2/13 | 1/4 | 0/16 | 2/8 | 2/16 | 0/1 | 0/6 | 0/11 | 1/20 | 1/2 | 0/19
Serious Adverse Events (participants affected / at risk) | 2/4 | 0/3 | 1/3 | 0/3 | 2/7 | 4/7 | 1/3 | 2/3 | 5/13 | 3/4 | 9/16 | 6/8 | 5/16 | 1/1 | 2/6 | 4/11 | 11/20 | 2/2 | 8/19
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3 | 3/3 | 3/3 | 7/7 | 7/7 | 3/3 | 3/3 | 12/13 | 4/4 | 16/16 | 8/8 | 16/16 | 1/1 | 6/6 | 11/11 | 19/20 | 2/2 | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Q2D Dose Escalation Phase: TAK-580 20 mg (22 Days Cycle) (N=4) | Q2D Dose Escalation Phase: TAK-580 40 mg (22 Days Cycle) (N=3) | Q2D Dose Escalation Phase: TAK-580 80 mg (22 Days Cycle) (N=3) | Q2D Dose Escalation Phase: TAK-580 135 mg (22 Days Cycle) (N=3) | Q2D Dose Escalation Phase: TAK-580 200 mg (22 Days Cycle) (N=7) | Q2D Dose Escalation Phase: TAK-580 280 mg (22 Days Cycle) (N=7) | Q2D Dose Escalation Phase: TAK-580 200 mg (28 Days Cycle) (N=3) | QW Dose Escalation Phase: TAK-580 400 mg (28 Days Cycle) (N=3) | QW Dose Escalation Phase: TAK-580 600 mg (28 Days Cycle) (N=13) | QW Dose Escalation Phase: TAK-580 800 mg (28 Days Cycle) (N=4) | Q2D Dose Expansion Phase: TAK-580 (BRAF+ Naive) (N=16) | Q2D Dose Expansion Phase: TAK-580 (BRAF+ Previously Treated) (N=8) | Q2D Dose Expansion Phase: TAK-580 (NRAS+ Naive) (N=16) | Q2D Dose Expansion Phase: TAK-580 (NRAS+ Previously Treated) (N=1) | Q2D Dose Expansion Phase: TAK-580 BRAF/NRAS WT+ Naive (N=6) | Q2D Dose Expansion Phase:TAK-580 BRAF/NRASWT+PreviouslyTreated (N=11) | Q2D Dose Expansion Phase: Pharmacokinetic Cohort (N=20) | Q2D Dose Expansion Phase: TAK-580 (BRAF+) (N=2) | QW Dose Expansion Phase: TAK-580 NRAS WT+ Naive (N=19)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (11) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticular perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Escherichia sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adverse drug reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Guillain-Barre syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ejection fraction decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Q2D Dose Escalation Phase: TAK-580 20 mg (22 Days Cycle) (N=4) | Q2D Dose Escalation Phase: TAK-580 40 mg (22 Days Cycle) (N=3) | Q2D Dose Escalation Phase: TAK-580 80 mg (22 Days Cycle) (N=3) | Q2D Dose Escalation Phase: TAK-580 135 mg (22 Days Cycle) (N=3) | Q2D Dose Escalation Phase: TAK-580 200 mg (22 Days Cycle) (N=7) | Q2D Dose Escalation Phase: TAK-580 280 mg (22 Days Cycle) (N=7) | Q2D Dose Escalation Phase: TAK-580 200 mg (28 Days Cycle) (N=3) | QW Dose Escalation Phase: TAK-580 400 mg (28 Days Cycle) (N=3) | QW Dose Escalation Phase: TAK-580 600 mg (28 Days Cycle) (N=13) | QW Dose Escalation Phase: TAK-580 800 mg (28 Days Cycle) (N=4) | Q2D Dose Expansion Phase: TAK-580 (BRAF+ Naive) (N=16) | Q2D Dose Expansion Phase: TAK-580 (BRAF+ Previously Treated) (N=8) | Q2D Dose Expansion Phase: TAK-580 (NRAS+ Naive) (N=16) | Q2D Dose Expansion Phase: TAK-580 (NRAS+ Previously Treated) (N=1) | Q2D Dose Expansion Phase: TAK-580 BRAF/NRAS WT+ Naive (N=6) | Q2D Dose Expansion Phase:TAK-580 BRAF/NRASWT+PreviouslyTreated (N=11) | Q2D Dose Expansion Phase: Pharmacokinetic Cohort (N=20) | Q2D Dose Expansion Phase: TAK-580 (BRAF+) (N=2) | QW Dose Expansion Phase: TAK-580 NRAS WT+ Naive (N=19)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 12 (42) | 7 (23) | 9 (11) | 0 (0) | 3 (3) | 1 (1) | 6 (10) | 0 (0) | 4 (5)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 5 (5) | 1 (1) | 5 (5) | 1 (1) | 5 (5) | 0 (0) | 1 (1) | 1 (2) | 11 (15) | 2 (2) | 5 (6)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (4) | 2 (3) | 0 (0) | 0 (0) | 2 (5) | 1 (1) | 2 (5) | 3 (3) | 4 (9) | 1 (2) | 3 (4)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 3 (4) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 5 (6) | 0 (0) | 1 (4)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 2 (3) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 3 (5) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (3)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retching (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip swelling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chapped lips (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glossodynia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip dry (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Salivary gland pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 3 (3) | 1 (1) | 1 (1) | 2 (2) | 6 (8) | 6 (7) | 1 (1) | 3 (3) | 6 (7) | 2 (2) | 5 (5) | 3 (4) | 7 (8) | 0 (0) | 3 (4) | 3 (3) | 12 (13) | 1 (1) | 9 (12)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 3 (5) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 7 (9) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (5) | 0 (0) | 7 (9) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 3 (4)
Face oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Localised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Axillary pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling cold (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site bruising (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 4 (5) | 2 (3) | 0 (0) | 2 (2) | 0 (0) | 7 (11) | 3 (5) | 9 (18) | 0 (0) | 1 (1) | 2 (2) | 7 (9) | 0 (0) | 2 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 3 (4) | 4 (4) | 0 (0) | 2 (3) | 1 (1) | 4 (5) | 0 (0) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (8) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 2 (3) | 3 (3) | 0 (0) | 2 (2)
Hair colour changes (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (7) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 2 (2)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (8) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 2 (3) | 1 (4) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Madarosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin mass (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitiligo (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Butterfly rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertrichosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Livedo reticularis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin plaque (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 1 (3) | 3 (3) | 0 (0) | 2 (2) | 2 (2) | 9 (9) | 1 (1) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 4 (4) | 0 (0) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (4) | 2 (3) | 3 (3) | 1 (1) | 2 (3) | 3 (5) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 1 (3) | 3 (4) | 3 (3) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 1 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 8 (13) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 5 (7) | 6 (10) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 4 (4) | 0 (0) | 1 (2) | 2 (3) | 5 (8) | 2 (2) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (2) | 3 (3) | 2 (2) | 0 (0) | 2 (2)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 2 (6)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 4 (7) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Blood calcium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood phosphorus decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Blood sodium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Blood folate decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood potassium increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breath sounds abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram T wave inversion (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 0 (0) | 4 (5) | 2 (2) | 1 (2) | 0 (0) | 2 (5) | 0 (0) | 2 (2) | 0 (0) | 2 (3)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 3 (4) | 3 (3) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Ageusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nervous system disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Poor quality sleep (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 6 (8) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 2 (2) | 9 (10) | 1 (1) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 5 (5) | 0 (0) | 2 (2)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Restrictive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 2 (2) | 4 (5) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 4 (5)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 3 (4) | 2 (2) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 1 (1) | 4 (4) | 3 (3) | 5 (7) | 2 (2) | 7 (9) | 1 (1) | 1 (1) | 5 (9) | 9 (13) | 2 (2) | 4 (5)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Reticulocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tinea infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biliary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear lobe infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Genital infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Klebsiella bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periorbital oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 3 (4) | 1 (1) | 2 (3)
Eye swelling (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelash discolouration (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (19) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye pruritus (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eyelid disorder (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelid irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelids pruritus (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Optic nerve disorder (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scleral haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitreous floaters (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral coldness (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Raynaud's phenomenon (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vena cava thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ureteric obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (6)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mood altered (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctival abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stoma site pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Metastases to chest wall (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear disorder (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Motion sickness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrophic vulvovaginitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast oedema (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scrotal oedema (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Statistical Analysis Plan (2016-07-29): https://cdn.clinicaltrials.gov/large-docs/08/NCT01425008/SAP_000.pdf
  • Study Protocol (2017-05-16): https://cdn.clinicaltrials.gov/large-docs/08/NCT01425008/Prot_001.pdf